CLINICAL TRIAL: NCT01828658
Title: Bioimpedance Versus Clinical Methods in Guiding Ultrafiltration in Hemodialysis Patients: a Randomized Trial
Brief Title: Randomized Bioimpedance vs Clinical Methods in Guiding Ultrafiltration in Hemodialysis Patients
Acronym: BIAHD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Grigore T. Popa University of Medicine and Pharmacy (Other)
Responsible Party: Principal Investigator, Professor Adrian Covic, Professor Dr., Grigore T. Popa University of Medicine and Pharmacy
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BCM0913
Record Dates: First submitted 2013-04-07; First posted 2013-04-10 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Haemodialyzed Patients; Volume Status
Keywords: hemodialysis; fluid management; bioimpedance; mortality; arterial stiffness

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Clinical (control) (No Intervention): In the clinical arm, dry weight and ultrafiltration prescription were done exclusively using traditional clinical methods of volume assessment.
- Bioimpedance arm (Active Comparator): Strict bioimpedance guided dry weight prescription arm. All patients dry weights were permanently maintained in the dry weight interval recommended by the BCM device (+/- 1,1 kg); BCM measurements were performed every 3 months.
  Interventions: Other: Strict bioimpedance guided dry weight prescription

INTERVENTIONS:
Other: Strict bioimpedance guided dry weight prescription — Post dialysis patient dry weight was exclusively prescribed using the ideal weight measured by the BCM device (+/- 1.1 Kg).
  Arms: Bioimpedance arm

SUMMARY:
The investigators developed a prospective, randomized, controlled trial to compare strict volume control using bioimpedance (using the BCM - Body Composition Monitor device) versus traditional clinical volume control in hemodialysis patients and the impact on mortality, hydration status, blood pressure values and arterial stiffness.

DETAILED DESCRIPTION:
The investigators developed a randomized controlled study to compare exclusively bioimpedance guided ultrafiltration in hemodialysis patients versus traditional methods for volume assessment.

The duration of the study was 3,5 years.

During the first 2,5 years of the study all enrolled patients were randomized using a block randomization algorithm in two arms.

In the interventional arm the post-dialysis dry weight was prescribed exclusively using the BCM device (Body Composition Monitor - Fresenius Medical Care, Germany).

In the control arm dry weight assessment was done by traditional clinical methods.

In both arms,during the intervention period (2,5 years) BCM measurements were performed every 3 months before dialysis, but only in the interventional arm the values were disclosed to the medical personnel and used to guide the dry weight and ultrafiltration volumes.

In the control arm (clinical), both patients and caregivers were fully blinded from the BCM results.

The BCM device measures for each patient an ideal dry weight interval ( +/- 1.1 kg). In the interventional arm, the prescribed dry weights of the patients were strictly maintained in the ideal weight interval (+/- 1.1 kg) proposed by the BCM device.

Primary outcome was all cause-mortality compared in the strict bioimpedance arm versus the clinical (control) arm and was assessed at 2,5 years.

Secondary end-points, assessed during the randomization period (2,5 years), were to compare blood pressure (determined pre dialysis), arterial stiffness and relative fluid overload (RFO = overhydration/ total body water), as measured by the BCM device.

During the last year of the study, all patients were left free of any intervention, and only arterial stiffness was assessed a third time at 3,5 years.

ELIGIBILITY:
Inclusion Criteria:

* older than 18-year
* on chronic hemodialysis for more than 3 months

Exclusion Criteria:

- life expectancy of less than 1 year

Presence of a condition that may interfere with the determination of dry weight using the Body Composition Monitor (R):

* severe ascites (decompensated liver failure)
* limb amputations
* cardiac stent, pacemaker or defibrillator
* hip prosthetic
* pregnancy
* mental deficiency (impossibility to give consent)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2008-07; Primary Completion 2010-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 2,5 years follow-up
  We assessed all-cause mortality in the two arms of the study at the end of intervention period.

SECONDARY OUTCOMES:
Arterial stiffness | 3,5 years
  Arterial stiffness was evaluated by applanation tonometry, measuring pulse wave velocity, and was done with a SphygmoCor® device (AtCor Medical, Westmead, Sydney, Australia).
  Measurements were performed in both arms at baseline, end of intervention (2,5 years) and at the end of the study (3,5 years).
Blood pressure values | 2,5 years
  In both arms, blood pressure was measured predialysis every 3 months and noted as a mean of the previous 3 predialysis BP values.
Overhydration | 2,5 years
  Overhydration was evaluated in both arms of the study using the Body Composition Monitor (BCM device), every 3 months. Overhydration was quantified as Relative fluid overload (RFO = overhydration/ total body water - as measured by the BCM.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Covic, Professor, Principal Investigator — University of Medicine and Pharmacy Iasi, "Dr. C.I.Parhon" University Hospital Iasi, Nephrology Department

REFERENCES:
- [Derived] Onofriescu M, Hogas S, Voroneanu L, Apetrii M, Nistor I, Kanbay M, Covic AC. Bioimpedance-guided fluid management in maintenance hemodialysis: a pilot randomized controlled trial. Am J Kidney Dis. 2014 Jul;64(1):111-8. doi: 10.1053/j.ajkd.2014.01.420. Epub 2014 Feb 28. PMID 24583055